CLINICAL TRIAL: NCT04373083
Title: Anti-PD-1 Antibody Treatment With Cemiplimab and Radiotherapy in Early-stage Favorable Classical Hodgkin Lymphoma (CARHL) - A Randomized Phase II Trial
Brief Title: Anti-PD-1 Antibody Treatment With Cemiplimab and Radiotherapy in Early-stage Classical Hodgkin Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R2810-ONC-1615; 2017-004265-28 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-05-04 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Hodgkin Lymphoma
Keywords: Early Stage; Favorable; Classical; classical Hodgkin lymphoma (cHL)
MeSH Terms: conditions — Hodgkin Disease | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Concomitant treatment (Experimental): Treatment Group A
  Interventions: Drug: Cemiplimab; Radiation: Involved-site radiotherapy (IS-RT)
- Sequential treatment (Experimental): Treatment Group B
  Interventions: Drug: Cemiplimab; Radiation: Involved-site radiotherapy (IS-RT)

INTERVENTIONS:
Drug: Cemiplimab — Administered in 3-week intervals
  Other Names: REGN2810; Libtayo
Radiation: Involved-site radiotherapy (IS-RT) — Patients will receive IS-RT with a dose of 20 Gy. Involved-site radiotherapy will be carried out on the basis of 3D imaging as described in the protocol

SUMMARY:
The primary objective is to estimate the efficacy of experimental treatment with the anti-PD-1 antibody cemiplimab (REGN2810) in combination with simultaneous or subsequent radiotherapy (RT) in early-stage favorable classical Hodgkin lymphoma (cHL).

Secondary objectives are to assess the safety and feasibility of the 2 experimental strategies.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically proven classical HL
* First diagnosis, no previous treatment
* Stage I-II without risk factors as defined in the protocol

Key Exclusion Criteria:

* Composite lymphoma or nodular lymphocyte-predominant Hodgkin lymphoma (NLPHL)
* Prior malignancy within the previous 5 years (except for locally treatable cancers that have been apparently cured by complete resection)
* Prior chemotherapy or radiation therapy
* Concurrent disease precluding protocol treatment as defined in the protocol
* Pregnancy or breast-feeding
* Non-compliance as defined in the protocol

Note: Other protocol-defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-15 (Estimated); Primary Completion 2022-12-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) at 1 year | From randomization up to 1 year

SECONDARY OUTCOMES:
PFS at 2 and 3 years | From randomization up to 3 years
Overall survival (OS) at 1, 2, and 3 years | From randomization up to 3 years
Incidence of acute toxicities | Up to 90 days after study treatment
Rate of patients with long-term fatigue using EORTC-QLQ-FA12 | 12-18 months after randomization
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ).
  -FA12 module complements the core EORTC QLQ-C30 questionnaire regarding fatigue. Each item can be scored in four dimension on a scale from 1 to 4 with higher scores indicating worse symptoms.
Rate of patients with long-term fatigue using EORTC-QLQ-C30 | 12-18 months after randomization
  Scores range from 0 to 100. A high scale score represents a higher response level.
Quality of life (QoL) using EORTC-QLQ-30 | Up to 3 years
  Scores range from 0 to 100. A high scale score represents a higher response level.
Rate of early discontinuation of study treatment | From first dose to up to 19 weeks
Frequency of lymphoma treatment administered in addition to study treatment | From randomization up to 3 years
Types of lymphoma treatment administered in addition to study treatment | From randomization up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/